CLINICAL TRIAL: NCT01928472
Title: Phase I Multi-center, Observer-Blind, Randomized Dose-Ranging Study of Adjuvanted and Non-Adjuvanted Cell Culture-Derived, Inactivated A/H7N9 Monovalent Subunit Influenza Virus Vaccine (H7N9c) in Adults 18 to <65 Years
Brief Title: Dose-finding Study of Four Dosage Levels of an H7N9 Influenza Vaccine in Adults Between Ages of 18 Years and 65 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Vaccines (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: V131_01
Record Dates: First submitted 2013-08-21; First posted 2013-08-26 (Estimated); Results first posted 2015-05-21 (Estimated); Last update posted 2019-06-11 (Actual); Status verified 2019-05

CONDITIONS: H7N9 Influenza
Keywords: Influenza, H7N9, Vaccine
MeSH Terms: conditions — Influenza, Human; Influenza in Birds | interventions — Adjuvants, Pharmaceutic

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- Group A (Experimental): H7N9c low dose with adjuvant
  Interventions: Biological: H7N9c low dose with adjuvant
- Group B (Experimental): H7N9c medium dose with adjuvant
  Interventions: Biological: H7N9c medium dose with adjuvant
- Group C (Experimental): H7N9c high dose with adjuvant
  Interventions: Biological: H7N9c high dose with adjuvant
- Group D (Experimental): H7N9c high dose without adjuvant
  Interventions: Biological: H7N9c high dose without adjuvant

INTERVENTIONS:
Biological: H7N9c low dose with adjuvant
  Arms: Group A
Biological: H7N9c medium dose with adjuvant
  Arms: Group B
Biological: H7N9c high dose with adjuvant
  Arms: Group C
Biological: H7N9c high dose without adjuvant
  Arms: Group D

SUMMARY:
Evaluate the safety and immunogenicity of four different doses of H7N9 vaccination in adults between the ages of 18 years and 65 years.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult subject ages 18-64 years.
2. Individuals willing to provide written informed consent
3. Individuals in good health.
4. Individuals who can comply with study procedures and follow-up.

Exclusion Criteria:

1. Individuals with history of cognitive or behavioral impairment or psychiatric disease,
2. Individuals unable to understand and follow study procedures,
3. History of significant illness,
4. History of chronic medical condition or progressive disease,
5. Allergy to any vaccine component or adverse event related to a vaccine component,
6. Impairment/alteration of the immune system,
7. Presence of progressive or severe neurological disorder,
8. Pregnant or breast-feeding,
9. Female of Child-bearing potential unwilling to use acceptable method of birth control,
10. Presence of medically significant cancer,
11. Receipt of investigational product within 30 day prior to entry into the study,
12. History of previous or suspected illness from avian flu caused by H7N9 virus,
13. History of H7 vaccination,
14. Body temperature of greater than or equal to 38.0°C (100.4◦F) and/or acute illness within 3 days of intended study vaccination,
15. Receipt of any flu vaccination 2 weeks before study entry or 4 weeks after study vaccination,
16. Receipt of any vaccination 2 weeks before study entry or 4 weeks after study vaccination,
17. History of drug or alcohol abuse within the past 2 years,
18. Body Mass Index (BMI) greater than or equal to 35kg/m2,
19. Individuals conducting the study or their immediate family members.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 402 (Actual)
Dates: Start 2013-08; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Vaccines and Diagnostics, Study Chair — Novartis Vaccines
Locations (6):
- United States (6):
  - Site 04: Accelovance, San Diego, California
  - Site 01: Accelovance, Melbourne, Florida
  - Site 02: Accelovance, Peoria, Illinois
  - Site 03: Accelovance, Rockville, Maryland
  - Site 05: Janet Lewis, Salt Lake City, Utah
  - Site 06: Janet Lewis, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 6 centers in United States.
Pre-assignment Details: All enrolled subjects were included in the trial.
Groups:
- Low Dose + Adj; Medium Dose + Adj; High Dose + Adj: Subjects received two doses of MF59 adjuvanted H7N9c vaccine formulation, administered three weeks apart
- High Dose + No Adj: Subjects received two doses of unadjuvanted of H7N9c vaccine formulation, administered three weeks apart.
Period: Overall Study
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Started | 98 | 104 | 98 | 102
Completed | 90 | 96 | 91 | 100
Not Completed | 8 | 8 | 7 | 2
Not completed — Death | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 4 | 1 | 2
Not completed — Lost to Follow-up | 2 | 3 | 4 | 0
Not completed — Administrative Reason | 2 | 1 | 0 | 0
Not completed — Unclassified | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- TOTAL: Total of all reporting groups
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj | TOTAL
Number analyzed (Participants) | 98 | 104 | 98 | 102 | 402
Age, Continuous [Mean (Standard Deviation); unit: year] | 38.3 (13.1) | 40.3 (12.5) | 42.6 (13.1) | 43.4 (12.9) | 41.2 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  FEMALE | 60 | 57 | 48 | 53 | 218
  MALE | 38 | 47 | 50 | 49 | 184

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers Of Subjects After Each Vaccination Of a Cell-Culture Derived H7N9c Monovalent Vaccine, Hemagglutination Inhibition Assay (Day 43)
Description: Immunogenicity was measured by Hemagglutination Inhibition (HI) assay and summarized through the geometric mean titers (GMTs) at baseline (day 1) and three weeks after the second (day 43) vaccination
Time Frame: Day 1 and 43
Population: The analysis was done on Full Analysis Set - Subjects who received at least one study vaccination and provided immunogenicity at day 43 (FAS-Day 43).
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
Titers
  Day 1 | 5 [4.95 to 5.05] | 5 [4.95 to 5.05] | 5 [4.95 to 5.05] | 5.05 [5 to 5.1]
  Day 43: number analyzed (Participants) | 94 | 103 | 97 | 102
  Day 43 | 12 [9.75 to 15] | 19 [15 to 23] | 26 [21 to 32] | 5.75 [4.67 to 7.08]

2. Primary Outcome: Geometric Mean Ratios In Subjects After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine, HI Assay (Day 43)
Description: Geometric mean ratio (GMR) of subjects was calculated as the ratio of postvaccination to prevaccination HI GMTs three weeks after second (day 43) vaccination.
Time Frame: Day 43
Population: FAS-Day 43
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 94 | 103 | 97 | 102
Ratio | 2.42 [1.95 to 3] | 3.7 [3.02 to 4.55] | 5.2 [4.21 to 6.43] | 1.14 [0.93 to 1.4]

3. Primary Outcome: Percentages Of Subjects Achieving Seroconversion After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Day 43)
Description: Percentage of subjects achieving HI seroconversion in HI titer was measured three weeks after second (day 43) vaccination.
  Seroconversion is defined as postvaccination HI titer> 40 for subjects with baseline (day 1); HI titer <1:10 or a minimum 4-fold increase in titer for subjects with baseline titer >1:10.
Time Frame: Day 43
Population: FAS-Day 43
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 94 | 103 | 97 | 102
Percentages of subjects | 26 [17 to 36] | 44 [34 to 54] | 52 [41 to 62] | 3 [1 to 8]

4. Primary Outcome: Percentages Of Subjects With an HI Titers ≥1:40 After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Day 43)
Description: Percentage of subjects who achieved HI titers≥1:40 was measured at baseline (day 1) and three weeks after second (Day 43) vaccination.
Time Frame: Day 1 and 43
Population: FAS-Day 43.
Measure: Number (95% Confidence Interval); unit: Percentages of subejcts
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
Percentages of subejcts
  Day 1 | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4]
  Day 43: number analyzed (Participants) | 94 | 103 | 97 | 102
  Day 43 | 26 [17 to 36] | 44 [34 to 54] | 52 [41 to 62] | 3 [1 to 8]

5. Secondary Outcome: Geometric Mean Titers Of Subjects After Each Vaccination Of A Cell-Culture Derived H7N9c Monovalent Vaccine, HI Assay (Day 22)
Description: Immunogenicity was measured by HI assay and summarized through the GMTs at baseline (day 1) and three weeks after the first (day 22) vaccination.
Time Frame: Day 1 and 22
Population: FAS-Day 22
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
Titers
  Day 1 | 5 [4.95 to 5.05] | 5 [4.95 to 5.05] | 5 [4.95 to 5.05] | 5.05 [5 to 5.1]
  Day 22 (N=96,103,97,102): number analyzed (Participants) | 96 | 103 | 97 | 102
  Day 22 (N=96,103,97,102) | 5.07 [4.95 to 5.2] | 5 [4.88 to 5.12] | 5 [4.88 to 5.13] | 5.1 [4.98 to 5.23]

6. Secondary Outcome: Geometric Mean Ratios In Subjects After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine, HI Assay (Day 22)
Description: GMR of subjects was calculated as the ratio of postvaccination to prevaccination HI GMTs three weeks after first (day 22) vaccination.
Time Frame: Day 22
Population: FAS-Day 22
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 96 | 103 | 97 | 102
Ratio | 1.01 [1 to 1.03] | 1 [0.98 to 1.02] | 1 [0.98 to 1.02] | 1.01 [0.99 to 1.03]

7. Secondary Outcome: Percentages Of Subjects Achieving Seroconversion After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Day 22)
Description: Percentage of subjects achieving HI seroconversion in HI titer was measured three weeks after first (day 22) vaccination.
  Seroconversion is defined as postvaccination HI titer> 40 for subjects with baseline (day 1); HI titer <1:10 or a minimum 4-fold increase in titer for subjects with baseline titer >1:10.
Time Frame: Day 22
Population: FAS-Day 22
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 96 | 103 | 97 | 102
Percentages of subjects | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4]

8. Secondary Outcome: Percentages Of Subjects With an HI Titers≥1:40 After Each Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Day 22)
Description: Percentage of subjects who achieved HI titers≥1:40 was measured at baseline (day 1) and three weeks after first (Day 22) vaccination.
Time Frame: Day 1 and 22.
Population: FAS-Day 22
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
Percentages of subjects
  Day 1 | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4]
  Day 22 | 0 [0 to 4] | 0 [0 to 4] | 0 [0 to 4] | 1 [0.025 to 5]

9. Secondary Outcome: Geometric Mean Titers at Six Months and One Year After Vaccination Of A Cell-Culture Derived H7N9c Vaccine, HI Assay (Persistence)
Description: The immunogenicity was measured as GMTs in subjects as persistence at six months (day 183) and one year (day 366) after the first vaccination as measured by Hemagglutination Inhibition (HI) Assay.
Time Frame: Day 183 and 366.
Population: FAS-Day 183 and FAS-Day 366
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 90 | 101 | 94 | 101
Titers
  Day 183 | 5.17 [4.84 to 5.52] | 5.43 [5.1 to 5.78] | 5.99 [5.61 to 6.39] | 5.16 [4.84 to 5.49]
  Day 366 (N=90,96,91,100): number analyzed (Participants) | 90 | 96 | 91 | 100
  Day 366 (N=90,96,91,100) | 5 [4.78 to 5.23] | 5.14 [4.92 to 5.37] | 5.14 [4.92 to 5.38] | 5.16 [4.94 to 5.38]

10. Secondary Outcome: Geometric Mean Ratios at Six Months and One Year After the First Vaccination Of A Cell-Culture Derived H7N9c Vaccine, HI Assay (Persistence)
Description: GMR of subjects was calculated as the ratio of postvaccination to prevaccination HI GMTs six months (day 183) and one year (day 366) after the first vaccination.
Time Frame: Day 183 and 366
Population: FAS-Day 183 and FAS-Day 366
Measure: Geometric Mean (95% Confidence Interval); unit: Ratio
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 90 | 101 | 94 | 101
Ratio
  Day 183/Day 1 | 1.03 [0.97 to 1.1] | 1.09 [1.02 to 1.15] | 1.2 [1.13 to 1.27] | 1.02 [0.96 to 1.08]
  Day 366/Day 1: number analyzed (Participants) | 90 | 96 | 91 | 100
  Day 366/Day 1 | 1 [0.96 to 1.04] | 1.03 [0.99 to 1.07] | 1.03 [0.99 to 1.07] | 1.02 [0.98 to 1.06]

11. Secondary Outcome: Percentages Of Subjects Achieving Seroconversion at Six Months and One Year After Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Persistence)
Description: Percentage of subjects with HI seroconversion was measured as HI titer persistence at six months (day 183) and one year (day 366) after the first vaccination.
  Seroconversion is defined as postvaccination HI titer>40 for subjects with baseline (day 1); HI titer <1:10 or a minimum four-fold increase in titer for subjects with baseline titer>1:10.
Time Frame: Day 183 and 366
Population: FAS-Day 183 and FAS-Day 366
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 90 | 101 | 94 | 101
Percentages of subjects
  Day 183 | 0 [0 to 4] | 1 [0.025 to 5] | 1 [0.027 to 6] | 1 [0.025 to 5]
  Day 366: number analyzed (Participants) | 90 | 96 | 91 | 100
  Day 366 | 0 [0 to 4] | 1 [0.026 to 6] | 0 [0 to 4] | 1 [0.025 to 5]

12. Secondary Outcome: Percentages Of Subjects With an HI Titers ≥1:40 at Six Months and at One Year After the First Vaccination Of A Cell-Culture Derived H7N9c Vaccine (Persistence)
Description: Percentages of subjects who achieved HI titers≥1:40 was measured at six months (day 183) and one year (day 366) after the first vaccination of a cell-culture derived H7N9 vaccine.
Time Frame: Day 183 and 366
Population: FAS-Day 183 and FAS-Day 366
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 90 | 101 | 94 | 101
Percentages of subjects
  Day 183 | 0 [0 to 4] | 1 [0.025 to 5] | 1 [0.027 to 6] | 1 [0.025 to 5]
  Day 366: number analyzed (Participants) | 90 | 96 | 91 | 100
  Day 366 | 0 [0 to 4] | 1 [0.026 to 6] | 0 [0 to 4] | 1 [0.025 to 5]

13. Primary Outcome: Number of Subjects Reporting Unsolicited Adverse Events After Receiving Adjuvanted and Unadjuvanted Formulations of H7N9c Vaccine
Description: Safety was assessed as the number of subjects who reported any AEs, and at least possibly related AEs are collected from day 1 to day 43 following vaccination with adjuvanted and unadjuvanted formulations of H7N9c vaccine.
Time Frame: Day 1 to Day 43
Population: Analysis was done on unsolicited safety set - All subjects in the exposed set with unsolicited AE data.
Measure: Number; unit: participants
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 97 | 103 | 98 | 102
participants
  Any AEs | 29 | 31 | 24 | 24
  At least possibly related AEs | 6 | 11 | 7 | 8

14. Primary Outcome: Number of Subjects Reporting Unsolicited Serious Adverse Events After Receiving Adjuvanted and Unadjuvanted Formulations of H7N9c Vaccine
Description: The number of subjects reporting unsolicited adverse events after receiving adjuvanted and unadjuvanted formulations of H7N9c vaccine was reported. Safety was assessed as the number of subjects who reported SAEs, at least possibly related SAEs, new onset of chronic diseases (NOCDs), medically attended AEs, AEs of Special Interest (AESIs), AEs leading to withdrawal from the study were collected from day 1 to day 366 following vaccination with adjuvanted and unadjuvanted formulations of H7N9 vaccine.
Time Frame: Day 1 to Day 366.
Population: Analysis was done on unsolicited safety set.
Measure: Number; unit: participants
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
participants
  SAEs | 2 | 2 | 3 | 1
  At least possibly related SAEs | 0 | 0 | 0 | 0
  AEs leading to withdrawal | 0 | 0 | 1 | 0
  Medically attended AE | 33 | 43 | 34 | 30
  AESI | 0 | 0 | 0 | 0
  NOCD | 1 | 7 | 5 | 3
  Death | 0 | 0 | 1 | 0

15. Primary Outcome: Number of Subjects Reporting Solicited Local and Systemic Adverse Events After Receiving Adjuvanted and Unadjuvanted Formulations of H7N9c Vaccine
Description: Safety was assessed as the number of subjects who reported solicited local and systemic adverse events from day 1 to day 7 of vaccination of adjuvanted and unadjuvanted formulations of H7N9c vaccine.
Time Frame: Day 1 through Day 7 after each vaccination.
Population: Analysis was done on the solicited safety set - All subjects in the exposed set with solicited AE data.
Measure: Number; unit: participants
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj
Number analyzed (Participants) | 98 | 103 | 98 | 102
participants
  Any local-Vaccination I | 47 | 77 | 60 | 30
  Vaccination I, Pain | 42 | 74 | 53 | 19
  Vaccination I, Ecchymosis | 2 | 2 | 2 | 5
  Vaccination I, Erythema | 11 | 16 | 13 | 11
  Vaccination I, Induration | 5 | 6 | 9 | 4
  Any systemic-Vaccination I | 40 | 56 | 44 | 42
  Vaccination I, Nausea | 11 | 12 | 8 | 5
  Vaccination I, Myalgia | 10 | 23 | 13 | 11
  Vaccination I, Arthralgia | 4 | 13 | 10 | 8
  Vaccination I, Headache | 23 | 36 | 23 | 20
  Vaccination I, Fatigue | 20 | 32 | 24 | 22
  Vaccination I, Vomiting | 3 | 2 | 2 | 0
  Vaccination I, Diarrhea | 10 | 9 | 6 | 7
  Vaccination I, Loss of appetite | 4 | 10 | 11 | 4
  Vaccination I, Malaise | 8 | 25 | 23 | 15
  Vaccination I,Body Temp (≥38°C) | 0 | 1 | 0 | 1
  Vaccination I, Prevention of pain and/or fever | 3 | 3 | 0 | 1
  Vaccination I, Treatment of pain and/or fever | 4 | 12 | 3 | 3
  Any Local-Vaccination II: number analyzed (Participants) | 95 | 102 | 97 | 102
  Any Local-Vaccination II | 39 | 58 | 46 | 27
  Vaccination II, Pain: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Pain | 34 | 53 | 45 | 21
  Vaccination II, Ecchymosis: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Ecchymosis | 1 | 3 | 0 | 4
  Vaccination II, Erythema: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Erythema | 11 | 12 | 6 | 9
  Vaccination II, Induration: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Induration | 9 | 16 | 4 | 6
  Any Systemic-Vaccination II (N=95,102,97,102): number analyzed (Participants) | 95 | 102 | 97 | 102
  Any Systemic-Vaccination II (N=95,102,97,102) | 33 | 37 | 33 | 25
  Vaccination II, Nausea: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Nausea | 10 | 9 | 9 | 7
  Vaccination II, Myalgia: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Myalgia | 8 | 16 | 14 | 7
  Vaccination II, Arthralgia: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Arthralgia | 5 | 12 | 12 | 3
  Vaccination II, Headache: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Headache | 18 | 19 | 17 | 11
  Vaccination II, Fatigue: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Fatigue | 13 | 19 | 15 | 15
  Vaccination II, Vomiting: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Vomiting | 1 | 0 | 1 | 1
  Vaccination II, Diarrhea: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Diarrhea | 5 | 6 | 4 | 8
  Vaccination II, Loss of appetite: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Loss of appetite | 4 | 10 | 7 | 6
  Vaccination II, Malaise: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Malaise | 8 | 17 | 14 | 9
  Vaccination II, Body Temp (≥38°C): number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Body Temp (≥38°C) | 0 | 2 | 0 | 0
  Vaccination II, Prevention of pain and/or fever: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Prevention of pain and/or fever | 0 | 1 | 0 | 1
  Vaccination II, Treatment of pain and (or)fever: number analyzed (Participants) | 95 | 102 | 97 | 102
  Vaccination II, Treatment of pain and (or)fever | 3 | 7 | 7 | 4

ADVERSE EVENTS:
Time Frame: Solicited and unsolicited AEs collected from Day 1 to Day 7; SAEs, NOCD, medically attended AEs, AEs leading to withdrawal, AESI and concomitant medications associated with these events are collected from day 1 through day 366.
Description: All Solicited AEs are classified as systematic assessment and all unsolicited AEs are classified as non-systematic assessment.
  Of total 402 subjects, 401 subjects received study vaccination and were included in the safety analysis. One subject withdrew consent to participate at visit 1 and did not receive any study vaccination
Arm/Group | Low Dose + Adj | Medium Dose + Adj | High Dose + Adj | High Dose + No Adj | TOTAL
Serious Adverse Events (participants affected / at risk) | 2/98 | 2/103 | 3/98 | 1/102 | 8/401
Other Adverse Events (participants affected / at risk) | 71/98 | 87/103 | 79/98 | 62/102 | 299/401
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose + Adj (N=98) | Medium Dose + Adj (N=103) | High Dose + Adj (N=98) | High Dose + No Adj (N=102) | TOTAL (N=401)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1 | 0 | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 0 | 1 | 0 | 1
APPENDICITIS (Infections and infestations) | 0 | 1 | 0 | 0 | 1
INFECTION (Infections and infestations) | 1 | 0 | 0 | 0 | 1
OSTEOMYELITIS (Infections and infestations) | 0 | 0 | 0 | 1 | 1
MULTIPLE FRACTURES (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 1
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 1
CEREBRAL INFARCTION (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 1
ASTHMA (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 1
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose + Adj (N=98) | Medium Dose + Adj (N=103) | High Dose + Adj (N=98) | High Dose + No Adj (N=102) | TOTAL (N=401)
DIARRHOEA (Gastrointestinal disorders) | 14 | 14 | 9 | 12 | 49
NAUSEA (Gastrointestinal disorders) | 18 | 19 | 13 | 9 | 59
VOMITING (Gastrointestinal disorders) | 5 | 4 | 3 | 1 | 13
FATIGUE (General disorders) | 26 | 36 | 32 | 30 | 124
INJECTION SITE INDURATION (General disorders) | 1 | 6 | 2 | 1 | 10
INJECTION SITE PAIN (General disorders) | 55 | 80 | 67 | 32 | 234
MALAISE (General disorders) | 15 | 32 | 29 | 20 | 96
NASOPHARYNGITIS (Infections and infestations) | 5 | 2 | 3 | 4 | 14
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 | 8 | 5 | 10 | 27
DECREASED APPETITE (Metabolism and nutrition disorders) | 7 | 17 | 14 | 10 | 48
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 11 | 28 | 21 | 11 | 71
MYALGIA (Musculoskeletal and connective tissue disorders) | 17 | 33 | 24 | 16 | 90
HEADACHE (Nervous system disorders) | 34 | 45 | 31 | 27 | 137

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days